CLINICAL TRIAL: NCT03651232
Title: Prenatal Yoga for Pregnancy Related Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P000344
Record Dates: First submitted 2018-07-09; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Yoga; Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga (Experimental): weekly prenatal yoga group class
  Interventions: Behavioral: yoga
- support (Active Comparator): weekly group support class
  Interventions: Behavioral: support group

INTERVENTIONS:
Behavioral: yoga — once weekly group yoga class for 12 weeks
  Arms: yoga
Behavioral: support group — once weekly group support class for 12 weeks
  Arms: support

SUMMARY:
This is a pilot feasibility study investigating prenatal yoga for pregnancy related back pain.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated pregnancies starting at 12-26 weeks of gestation
* pregnant women with and without back pain who had no regular yoga practice.

Exclusion Criteria:

* significant back pathology
* pregnancy complications
* non-English speaking
* otherwise were not able to participate (eg. transportation, scheduling issues)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
feasibility of recruitment | baseline
  recruitment rate

SECONDARY OUTCOMES:
back pain disability | baseline, 4, 8, 12 weeks
  Roland Morris Disability Questionnaire (range 0-24), lower better
back pain severity | baseline, 4, 8, 12 weeks
  Back Pain Severity Visual Analogue Scale (rage 0-10), lower better
pregnancy symptoms | baseline, 4, 8, 12 weeks
  Pregnancy Symptom Inventory (range 0-123), lower better
depression | baseline, 4, 8, 12 weeks
  Edinburgh Postnatal Depression Scale (range 0-30), lower better
quality of lfe | baseline, 4, 8, 12 weeks
  Short Form-12 (range 12-56), higher better
childbirth experience | postpartum visit
  Childbirth Experience (range 19-76), higher better
mobility lab- speed | baseline, 4, 8, 12 weeks
  instrumented gait speed
acceptability | 4,8, 12 weeks, postpartum
  class attendance
mobility lab- double support | baseline, 4, 8, 12 weeks
  double support time
mobility lab- TUG | baseline, 4, 8, 12 weeks
  timed up and go time
mobility lab- turn | baseline, 4, 8, 12 weeks
  turn time

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Yeh, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No